CLINICAL TRIAL: NCT04120116
Title: A Phase 2a, Prospective, Randomized, Double-Blind, Placebo-Controlled, Single and Repeat-Dose, Multicenter, Exploratory Efficacy Study of FX-322 Administered by Intratympanic Injection in Adults With Stable Sensorineural Hearing Loss
Brief Title: FX-322 in Adults With Stable Sensorineural Hearing Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Frequency Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FX-322-202
Record Dates: First submitted 2019-09-30; First posted 2019-10-09 (Actual); Results first posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Sensorineural Hearing Loss; Noise Induced Hearing Loss; Sudden Sensorineural Hearing Loss
Keywords: Intratympanic Administration; Restoration of Hearing Function
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss, Noise-Induced; Hearing Loss, Sudden

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- FX-322 Single Dose, Placebo Three Doses (Experimental): Four intratympanic injections of a hydrogel formulation, FX-322 Single Dose, Placebo Three Doses.
  Interventions: Drug: FX-322 (One Dose); Drug: Placebo
- FX-322 Two Doses, Placebo Two Doses (Experimental): Four intratympanic injections of a hydrogel formulation, FX-322 Two Doses, Placebo Two Doses.
  Interventions: Drug: FX-322 (Two Doses); Drug: Placebo
- FX-322 Four Doses (Experimental): Four intratympanic injections of a hydrogel formulation, FX-322 Four Doses.
  Interventions: Drug: FX-322 (Four Doses)
- Placebo Four Doses (Placebo Comparator): Four intratympanic injections of a hydrogel formulation, Placebo Four Doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FX-322 (One Dose) — Patients will receive one dose of FX-322.
  Arms: FX-322 Single Dose, Placebo Three Doses
Drug: FX-322 (Two Doses) — Patients will receive two doses of FX-322.
  Arms: FX-322 Two Doses, Placebo Two Doses
Drug: FX-322 (Four Doses) — Patients will receive four doses of FX-322.
  Arms: FX-322 Four Doses
Drug: Placebo — Patients will receive Placebo.
  Arms: FX-322 Single Dose, Placebo Three Doses; FX-322 Two Doses, Placebo Two Doses; Placebo Four Doses

SUMMARY:
This is a phase 2a single and repeat dose exploratory efficacy study of intratympanic FX-322 compared to placebo in healthy male and female adults with stable sensorineural hearing loss.

DETAILED DESCRIPTION:
Sensorineural hearing loss (SNHL) accounts for about 90% of all cases of hearing loss. This phase 2a study will assess the exploratory efficacy, as well as the local and systemic safety of single and repeat intratympanic doses of FX-322 compared to placebo in approximately 96 subjects with stable mild to moderately severe sensorineural hearing loss, with a medical history consistent with either excessive noise exposure or idiopathic sudden sensorineural hearing loss.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18-65 years inclusive.
2. Established diagnosis of stable sensorineural hearing loss by standard audiometric measures for ≥ 6 months prior to the Screening visit (no changes in air conduction greater than 10 dB at a single frequency or greater than 5 dB at two contiguous frequencies from the prior audiogram to the Screening audiogram in the study ear).
3. Documented medical history consistent with hearing loss being caused by noise exposure or sudden sensorineural hearing loss.
4. Pure Tone Audiometry (PTA) within 26-70 dB in the ear to be injected.
5. Female subjects must be of non-childbearing potential or will need to utilize two methods of highly effective contraception during the study participation (e.g. hormonal contraception or an intrauterine device and condoms) or remain abstinent. Male subjects should use condoms with spermicide during the course of the study or remain abstinent. Subjects should not donate sperm or ova during the study period.

Exclusion Criteria:

1. Previous participation in FX-322 clinical trial.
2. Currently on any medication consisting of valproic acid, valproate sodium, or divalproex sodium.
3. Perforation of tympanic membrane or other tympanic membrane disorders that would interfere with the delivery and safety assessment of an intratympanic medication or reasonably be suspected to affect tympanic membrane healing after injection in study ear. This includes a current tympanostomy tube.
4. Any conductive hearing loss of greater than 15 dB at a single frequency or greater than 10 dB at two or more contiguous octave frequencies in the study ear at the Screening visit or on the prior audiogram (if the Investigator feels there is not a true conductive hearing loss, the Medical Monitor should be consulted).
5. Active chronic middle ear disease or a history of major middle ear surgery, as an adult, in the ear to be injected.
6. Subject has had an intratympanic injection in either ear within 6 months of the screening visit.
7. History of clinically significant vestibular symptoms at the discretion of the investigator.
8. History of clinically significant systemic autoimmune disease.
9. History of head or neck radiation treatment or exposure.
10. History of platinum-based chemotherapy treatment.
11. Exposure to another investigational drug within 28 days prior to injection of study drug.
12. Evidence of any active or chronic disease or condition that could interfere with, or for which the treatment of might interfere with, the conduct of the study, or that would pose an unacceptable risk to the subject in the opinion of the investigator following a detailed medical history, physical examination, and vital signs (systolic and diastolic blood pressure, pulse rate, body temperature).
13. History of substance abuse within 2 years of the Screening Visit.
14. Positive test for drugs of abuse at screening.
15. Positive urine pregnancy test or breast-feeding.
16. Any known factor, condition or disease that, in the view of the Investigator, might interfere with treatment compliance, study conduct or interpretation of the results (e.g. previous high-dose aminoglycoside treatment).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2020-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl LeBel, PhD, Study Director — Frequency Therapeutics
Locations (15):
- United States (15):
  - Clinical Trial Site, Fresno, California
  - Clinical Trial Site, Torrance, California
  - Clinical Trial Site, Colorado Springs, Colorado
  - Clinical Trial Site, Boca Raton, Florida
  - Clinical Trial Site, Sarasota, Florida
  - Clinical Trial Site, Tampa, Florida
  - Clinical Trial Site, Louisville, Kentucky
  - Clinical Trial Site, Omaha, Nebraska
  - Clinical Trial Site, Amherst, New York
  - Clinical Trial Site, Matthews, North Carolina
  - Clinical Trial Site, Winston-Salem, North Carolina
  - Clinical Trial Site, Orangeburg, South Carolina
  - Clinical Trial Site, Austin, Texas
  - Clinical Trial Site, San Antonio, Texas
  - Clinical Trial Site, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: FX-322 Single Dose, Placebo Three Doses: Four weekly intratympanic injections:
  One dose of FX-322 (laduviglusib 0.628 mg/sodium valproate 17.72 mg) followed by three doses of placebo
- Group 2: FX-322 Two Doses, Placebo Two Doses: Four weekly intratympanic injections:
  Two doses of FX-322 (laduviglusib 0.628 mg/sodium valproate 17.72 mg) followed by two doses of placebo
- Group 3: FX-322 Four Doses: Four weekly intratympanic injections of FX-322 (laduviglusib 0.628 mg/sodium valproate 17.72 mg)
- Group 4: Placebo Four Doses: Four weekly intratympanic injections of placebo
Period: Overall Study
Arm/Group | Group 1: FX-322 Single Dose, Placebo Three Doses | Group 2: FX-322 Two Doses, Placebo Two Doses | Group 3: FX-322 Four Doses | Group 4: Placebo Four Doses
Started | 23 | 25 | 24 | 23
Completed | 22 | 24 | 22 | 20
Not Completed | 1 | 1 | 2 | 3
Not completed — Lost to Follow-up | 0 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1
Not completed — Subject was deemed to not meet the inclusion criteria for SNHL after dose was administered | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set is defined as all randomized subjects who received at least one dose of study drug or placebo in the study ear per the randomized treatment schedule
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: FX-322 Single Dose, Placebo Three Doses | Group 2: FX-322 Two Doses, Placebo Two Doses | Group 3: FX-322 Four Doses | Group 4: Placebo Four Doses | Total
Number analyzed (Participants) | 23 | 25 | 21 | 21 | 90
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.8 (8.93) | 54.4 (10.58) | 51.0 (13.61) | 55.1 (10.52) | 53.9 (10.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 3 | 7 | 26
  Male | 15 | 17 | 18 | 14 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 1 | 4 | 10
  Not Hispanic or Latino | 21 | 22 | 20 | 17 | 80
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 2 | 2 | 7
  White | 19 | 23 | 19 | 18 | 79
  More than one race | 1 | 1 | 0 | 0 | 2
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 23 | 25 | 21 | 21 | 90

OUTCOME MEASURES:

1. Primary Outcome: Word Recognition in Quiet
Description: Percent of subjects exceeding the Carney-Schlauch 95% confidence interval for improvement from baseline in number of words recognized from Consonant-Nucleus-Consonant (CNC) word lists
Time Frame: Baseline to Day 210
Population: Full Analysis Set is defined as all randomized subjects who received at least one dose of study drug or placebo in the study ear per the randomized treatment schedule. Only data from subjects in the FAS that attended the Day 210 visit were analyzed for this endpoint. The FX-322 Pooled Group consists of subjects in the Groups 1, 2, and 3 combined. The Pooled Group is for analysis only and does not signify a separate randomized group of subjects.
Measure: Number; unit: Percent
Groups:
- FX-322 Pooled: All participants (Groups 1, 2, and 3 combined) receiving at least one dose of FX-322 (laduviglusib 0.628 mg/sodium valproate 17.72 mg)
Arm/Group | Group 1: FX-322 Single Dose, Placebo Three Doses | Group 2: FX-322 Two Doses, Placebo Two Doses | Group 3: FX-322 Four Doses | FX-322 Pooled | Group 4: Placebo Four Doses
Number analyzed (Participants) | 21 | 24 | 19 | 64 | 17
Percent | 23.8 | 16.7 | 15.8 | 18.8 | 41.2
Statistical Analysis 1: Comparison: FX-322 Pooled vs Group 4: Placebo Four Doses; Test type: Superiority; p = 0.068, Mixed Models Analysis — P value for statistical significance is <0.05; Odds Ratio (OR) = 0.3, 95% CI 2-sided [0.11 to 1.08]

2. Primary Outcome: Words-in-Noise
Description: Mean absolute percent change in number of recognized words from CNC word lists
Time Frame: Baseline to Day 210
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Group 1: FX-322 Single Dose, Placebo Three Doses | Group 2: FX-322 Two Doses, Placebo Two Doses | Group 3: FX-322 Four Doses | FX-322 Pooled | Group 4: Placebo Four Doses
Number analyzed (Participants) | 21 | 24 | 19 | 64 | 17
Percent change | 2.58 (7.251) | 3.33 (8.933) | 1.80 (7.236) | 2.63 (7.822) | 3.61 (11.259)

3. Primary Outcome: Pure Tone Audiometry
Description: Mean overall pure tone average (PTA) hearing thresholds in decibels (dB) derived by averaging the air conduction thresholds at 0.5, 1, 2 and 4kHZ frequencies
Time Frame: Baseline to Day 210
Population: Full Analysis Set is defined as all randomized subjects who received at least one dose of study drug or placebo in the study ear per the randomized treatment schedule. Only data from subjects in the FAS that attended the Day 210 visit were analyzed for this endpoint. FX-322 Pooled Group consists of subjects in the Groups 1, 2, and 3 combined. The Pooled Group is for analysis only and does not signify a separate randomized group of subjects.
Measure: Least Squares Mean (Standard Error); unit: Decibels (dB)
Arm/Group | Group 1: FX-322 Single Dose, Placebo Three Doses | Group 2: FX-322 Two Doses, Placebo Two Doses | Group 3: FX-322 Four Doses | FX-322 Pooled | Group 4: Placebo Four Doses
Number analyzed (Participants) | 21 | 24 | 19 | 64 | 17
Decibels (dB) | 54.92 (2.284) | 55.08 (2.175) | 52.44 (2.372) | 54.15 (1.417) | 52.90 (2.404)
Statistical Analysis 1: Comparison: FX-322 Pooled vs Group 4: Placebo Four Doses; Test type: Superiority; p = 0.634, Mixed Models Analysis — P value for statistical significance is <0.05; Least squares mean difference = 1.25, 95% CI 2-sided [-3.945 to 6.439], Standard Error of Mean 2.611

4. Primary Outcome: Treatment-emergent Adverse Events (TEAEs)
Description: Number of patients with treatment-related adverse events assessed by CTCAE v5.0
Time Frame: Baseline to Day 210
Population: Safety Analysis Set (SAS) is defined as all subjects exposed to study drug or placebo. For TEAEs, subjects were analyzed per the treatment group that reflected the number of FX-322 doses actually administered. Two subjects who were initially randomized to Group 3 only received 3 of the 4 doses of FX-322 and were analyzed for TEAEs in the Total Group only. One subject who was initially randomized into Group 3 only received 1 of the 4 doses of FX-322 and therefore was analyzed in Group 1.
Measure: Count of Participants; unit: Participants
Groups:
- Total: Combination of Group 1, Group 2, Group 3, Group 4, and two subjects randomized to Group 3 who only received 3 of 4 doses of FX-322
Arm/Group | Group 1: FX-322 Single Dose, Placebo Three Doses | Group 2: FX-322 Two Doses, Placebo Two Doses | Group 3: FX-322 Four Doses | Group 4: Placebo Four Doses | Total
Number analyzed (Participants) | 24 | 25 | 21 | 23 | 95
Participants | 16 | 16 | 19 | 12 | 64

5. Primary Outcome: Otoscopy Abnormalities
Description: Number of treated ears with abnormalities of the external ear canal, tympanic membrane and middle ear at each specified time point
Time Frame: Baseline and Days 8, 15, 21 60, 90,150, and 210
Population: Safety Analysis Set (SAS) is defined as all subjects exposed to study drug or placebo. For otoscopies, subjects were analyzed per the treatment group that reflected the number of FX-322 doses actually administered. Two subjects who were initially randomized to Group 3 only received 3 of the 4 doses of FX-322 and were analyzed in the FX-322 Pooled Group only. One subject who was initially randomized into Group 3 only received 1 of the 4 doses of FX-322 and therefore was analyzed in Group 1.
Measure: Number; unit: Number of ears
Units Other Than Participants: Ears
Groups:
- FX-322 Pooled: Combination of Group 1, Group 2, Group 3, and two subjects randomized to Group 3 who only received 3 of 4 doses of FX-322.
Arm/Group | Group 1: FX-322 Single Dose, Placebo Three Doses | Group 2: FX-322 Two Doses, Placebo Two Doses | Group 3: FX-322 Four Doses | FX-322 Pooled | Group 4: Placebo Four Doses
Number analyzed (Participants) | 24 | 25 | 21 | 72 | 23
Number analyzed (Ears) | 24 | 25 | 21 | 72 | 23
Number of ears
  External - Baseline | 0 | 0 | 1 | 1 | 0
  External - Day 8 | 1 | 0 | 1 | 2 | 1
  External - Day 15 | 2 | 0 | 1 | 3 | 0
  External - Day 21 | 1 | 0 | 2 | 3 | 0
  External - Day 60 | 0 | 0 | 0 | 0 | 0
  External - Day 90 | 0 | 2 | 0 | 2 | 2
  External - Day 150 | 1 | 1 | 1 | 3 | 1
  External - Day 210 | 1 | 0 | 1 | 2 | 1
  Tympanic membrane - Baseline | 1 | 0 | 0 | 1 | 1
  Tympanic membrane - Day 8 | 2 | 3 | 1 | 7 | 2
  Tympanic membrane - Day 15 | 4 | 1 | 2 | 7 | 4
  Tympanic membrane - Day 21 | 2 | 1 | 3 | 6 | 1
  Tympanic membrane - Day 60 | 0 | 1 | 0 | 1 | 2
  Tympanic membrane - Day 90 | 0 | 1 | 0 | 1 | 2
  Tympanic membrane - Day 150 | 1 | 0 | 0 | 1 | 0
  Tympanic membrane - 210 | 0 | 0 | 0 | 0 | 1
  Middle Ear - Baseline | 0 | 0 | 0 | 0 | 0
  Middle Ear - Day 8 | 1 | 0 | 0 | 1 | 0
  Middle Ear - Day 15 | 1 | 0 | 1 | 2 | 1
  Middle Ear - Day 21 | 1 | 0 | 1 | 2 | 1
  Middle Ear - Day 60 | 0 | 0 | 0 | 0 | 0
  Middle Ear - Day 90 | 0 | 0 | 0 | 0 | 0
  Middle Ear - Day 150 | 0 | 0 | 0 | 0 | 0
  Middle Ear - Day 210 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Tympanometry Abnormalities
Description: Number of treated ears with changes in middle ear compliance (mL), peak pressure (daPa), and/or ear canal volume (mL) from baseline
Time Frame: Baseline and Days 15, 60, 90, 150, 210
Population: Safety Analysis Set (SAS) is defined as all subjects exposed to study drug or placebo. For tympanometry tests, subjects were analyzed per the treatment group that reflected the number of FX-322 doses actually administered. Two subjects who were initially randomized to Group 3 only received 3 of the 4 doses of FX-322 and were analyzed in the FX-322 Pooled Group only. One subject who was initially randomized into Group 3 only received 1 of the 4 doses of FX-322 and thus was analyzed in Group 1
Measure: Number; unit: Number of ears
Units Other Than Participants: Ears
Arm/Group | Group 1: FX-322 Single Dose, Placebo Three Doses | Group 2: FX-322 Two Doses, Placebo Two Doses | Group 3: FX-322 Four Doses | FX-322 Pooled | Group 4: Placebo Four Doses
Number analyzed (Participants) | 24 | 25 | 21 | 72 | 23
Number analyzed (Ears) | 24 | 25 | 21 | 72 | 23
Number of ears
  Baseline | 0 | 0 | 1 | 1 | 2
  Day 15 | 2 | 0 | 4 | 6 | 4
  Day 60 | 0 | 0 | 0 | 0 | 0
  Day 90 | 0 | 0 | 0 | 0 | 0
  Day 150 | 0 | 0 | 0 | 0 | 0
  Day 210 | 0 | 0 | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: Baseline through Day 210
Description: Safety Analysis Set (SAS) is defined as all subjects exposed to study drug or placebo. For AEs, subjects were analyzed per the treatment group that reflected the number of FX-322 doses actually administered. Two subjects who were initially randomized to Group 3 only received 3 of the 4 doses of FX-322 and were analyzed for AEs in the Total Group only. One subject who was initially randomized into Group 3 only received 1 of the 4 doses of FX-322 and therefore was analyzed in Group 1.
Arm/Group | Group 1: FX-322 Single Dose, Placebo Three Doses | Group 2: FX-322 Two Doses, Placebo Two Doses | Group 3: FX-322 Four Doses | Group 4: Placebo Four Doses | Total
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/25 | 0/21 | 0/23 | 0/95
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25 | 0/21 | 0/23 | 1/95
Other Adverse Events (participants affected / at risk) | 16/24 | 16/25 | 19/21 | 12/23 | 64/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: FX-322 Single Dose, Placebo Three Doses (N=24) | Group 2: FX-322 Two Doses, Placebo Two Doses (N=25) | Group 3: FX-322 Four Doses (N=21) | Group 4: Placebo Four Doses (N=23) | Total (N=95)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Deemed unrelated to study drug
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: FX-322 Single Dose, Placebo Three Doses (N=24) | Group 2: FX-322 Two Doses, Placebo Two Doses (N=25) | Group 3: FX-322 Four Doses (N=21) | Group 4: Placebo Four Doses (N=23) | Total (N=95)
Hypoacusis (Ear and labyrinth disorders) | 5 | 5 | 7 | 4 | 21
Ear discomfort (Ear and labyrinth disorders) | 3 | 2 | 6 | 1 | 12
Tinnitus (Ear and labyrinth disorders) | 5 | 3 | 1 | 0 | 9
Ear pain (Ear and labyrinth disorders) | 1 | 2 | 1 | 0 | 4
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1 | 1 | 3
Ear hemmorhage (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 2
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 2
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 2 | 0 | 2
Conductive deafness (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 1
Excessive cerumen production (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1
Otorrhea (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 1
Injection site pain (General disorders) | 2 | 3 | 3 | 2 | 10
Injection site scab (General disorders) | 0 | 1 | 1 | 3 | 5
Injection site hemorrhage (General disorders) | 2 | 1 | 0 | 1 | 4
Injection site discomfort (General disorders) | 0 | 0 | 2 | 0 | 2
Discomfort (General disorders) | 0 | 1 | 0 | 0 | 1
Facial pain (General disorders) | 0 | 1 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 1 | 2 | 5
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Eye infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Otitis externa fungal (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 1 | 3
Headache (Nervous system disorders) | 2 | 0 | 1 | 0 | 3
Balance disorder (Nervous system disorders) | 0 | 2 | 0 | 0 | 2
Dizziness postural (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Nystagmus (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Retinal migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Taste disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Visual field defect (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 2
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 2
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Audiogram abnormal (Investigations) | 0 | 1 | 1 | 1 | 3
Blood cholesterol increased (Investigations) | 1 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Nightmare (Psychiatric disorders) | 0 | 1 | 1 | 0 | 2
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 1 | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0 | 2
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Corneal irritation (Eye disorders) | 1 | 1 | 0 | 0 | 1
Glaucoma (Eye disorders) | 0 | 1 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hyperlipidemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs must obtain sponsor's written consent before publishing or presenting the trial results

DOCUMENTS (2):
  • Study Protocol (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/16/NCT04120116/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/16/NCT04120116/SAP_002.pdf